CLINICAL TRIAL: NCT07073742
Title: Randomized, Controlled, Non-Inferiority Trial on the Efficacy of CLaCS Using 0.2% Aetoxysklerol Foam and 70% Glucose for the Treatment of Lower Limb Telangiectasias
Brief Title: CLaCS Using 0.2% Aetoxysklerol Foam and 70% Glucose for the Treatment of Lower Limb Telangiectasias
Acronym: CLACSO
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 111111
Record Dates: First submitted 2025-07-10; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Varicose Veins of Lower Limb; Spider Veins; Reticular Leg Veins
Keywords: Telangiectasia; CryoLaser and CryoSclerotherapy; Cosmetic phlebology; AI prediction
MeSH Terms: conditions — Telangiectasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CLaCS with 70% Glucose (Control Group) (Active Comparator): Participants in this group will undergo the CLaCS procedure using Nd:YAG 1064 nm laser followed by intravascular injection of 70% glucose as the sclerosant. This represents the standard CLaCS protocol and serves as the control arm.
  Interventions: Procedure: CLaCS
- CLaCS with 0.2% Polidocanol Foam (Aetoxysklerol) - Test Group (Active Comparator): Participants in this group will receive the same laser treatment (Nd:YAG 1064 nm) as the control group, but the sclerosant will be a 0.2% polidocanol foam, prepared using the VARIXIO system. This arm evaluates the efficacy of a low-concentration detergent-based alternative.
  Interventions: Procedure: CLaCS

INTERVENTIONS:
Procedure: CLaCS — CLaCS is hybrid outpatient procedure combining Nd:YAG 1064 nm laser treatment with injection of a sclerosant (either 70% glucose or 0.2% polidocanol foam).

SUMMARY:
This randomized, controlled, non-inferiority trial aims to compare the efficacy of two sclerosants used in the CLaCS (CryoLaser and CryoSclerotherapy) method for treating telangiectasias and reticular varicose veins. CLaCS is an advanced outpatient procedure that combines Nd\:YAG laser treatment with sclerotherapy to enhance vein closure and cosmetic outcomes while minimizing side effects. The trial will compare the standard 70% glucose sclerosant with a novel 0.2% Aetoxysklerol (polidocanol) foam prepared using the VARIXIO system. Despite widespread use of CLaCS, no head-to-head studies currently exist comparing these two agents. This study aims to determine whether low-concentration Aetoxysklerol foam is non-inferior to 70% glucose in achieving effective telangiectasia elimination.

DETAILED DESCRIPTION:
Telangiectasias and reticular varicose veins affect up to 80% of the population, significantly impacting quality of life beyond cosmetic concerns. In advanced stages (e.g., corona phlebectatica), they may contribute to the progression of chronic venous disease. CLaCS (CryoLaser and CryoSclerotherapy) is currently regarded as the most advanced outpatient technique for managing these lesions. It integrates two modalities: laser-induced vasospasm of feeder veins using Nd:YAG 1064 nm laser, and subsequent sclerotherapy of the visible telangiectasias. This hybrid approach aims to maximize efficacy while minimizing adverse effects associated with each component when used in isolation.

The original CLaCS protocol utilizes 70% hypertonic glucose as the sclerosant, a substance that induces endothelial dehydration, fibrosis, and gradual obliteration of the treated veins. While glucose is widely considered safe and well tolerated, its efficacy may be limited in certain patient populations or lesion types.

Alternatively, polidocanol (Aetoxysklerol), a detergent-type sclerosant, is routinely used in concentrations of 0.5-3% for sclerotherapy. It disrupts the endothelial surface, triggering inflammation, spasm, and thrombosis, ultimately resulting in vessel closure. Recent advances in delivery techniques, such as the VARIXIO system, allow for the generation of a highly stable foam using very low concentrations of Aetoxysklerol (e.g., 0.2%). This approach may retain therapeutic efficacy while potentially reducing complications like hyperpigmentation, pain, or matting.

To date, no clinical trials have directly compared the effectiveness of CLaCS using different sclerosants. This prospective, randomized, controlled, non-inferiority trial aims to evaluate whether 0.2% Aetoxysklerol foam is non-inferior to 70% glucose in the treatment of lower limb telangiectasias using the CLaCS method. Patients will be randomly assigned to receive CLaCS treatment with either 70% glucose or 0.2% polidocanol foam, with outcomes assessed by blinded evaluators using standardized pre- and post-treatment photography and patient-reported satisfaction.

The primary endpoint is the proportion of treated areas showing clinically significant clearance of telangiectasias at 8 weeks post-treatment. Secondary endpoints include patient satisfaction and comparison of treatment outcomes with AI-based predictive modeling. This trial will provide critical evidence to inform sclerosant selection in CLaCS procedures and may support broader adoption of low-dose detergent-based foams as a safe and effective alternative to glucose.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Age > 18 years.
3. CEAP classification C1 (telangiectasias only).
4. Treated area for the study must be ≤ 20x20 cm on the lower limb - thigh.

Exclusion Criteria:

1. Reflux in trunk veins or perforators.
2. Active skin infection at the treatment site.
3. Presence of reticular veins.
4. Previous sclerotherapy/CLaCS in the target area.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 240 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
To assess the rate of telangiectasia elimination using CLaCS with two types of sclerosants (G-70 and AET-0.2). | 8 weeks

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bertanha M, Yoshida WB, Bueno de Camargo PA, Moura R, Reis de Paula D, Padovani CR, Sobreira ML. Polidocanol Plus Glucose Versus Glucose Alone for the Treatment of Telangiectasias: Triple Blind, Randomised Controlled Trial (PG3T). Eur J Vasc Endovasc Surg. 2021 Jan;61(1):128-135. doi: 10.1016/j.ejvs.2020.07.007. Epub 2020 Aug 7. PMID 32778489
- [Result] Miyake RK, Chi YW, Franklin IJ, Gianesini S. State of the art on cryo-laser cryo-sclerotherapy in lower limb venous aesthetic treatment. J Vasc Surg Venous Lymphat Disord. 2020 Sep;8(5):893-895. doi: 10.1016/j.jvsv.2020.01.003. Epub 2020 Mar 14. PMID 32179040
- [Result] Gonzalez Ochoa AJ, Carrillo J, Manriquez D, Manrique F, Vazquez AN. Reducing hyperpigmentation after sclerotherapy: A randomized clinical trial. J Vasc Surg Venous Lymphat Disord. 2021 Jan;9(1):154-162. doi: 10.1016/j.jvsv.2020.06.019. Epub 2020 Jul 30. PMID 32739509